CLINICAL TRIAL: NCT01915147
Title: A Study to Explore the Influence of Two Opioid Pain Medications on Bacterial Composition in the Gut and Other Gastrointestinal Aspects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OXN2505; 2012-001772-11 (EudraCT Number)
Record Dates: First submitted 2013-06-06; First posted 2013-08-02 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Severe Chronic Pain
Keywords: oxycodone naloxone combination; severe chronic pain; non-malignant pain; Non-malignant pain that requires around-the-clock opioid therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OXN PR followed by OxyPR tablets (Experimental): OXN PR followed by OxyPR tablets
  Interventions: Drug: OXN PR followed by OxyPR tablets
- OxyPR followed by OXN PR tablets (Experimental): OxyPR followed by OXN PR tablets
  Interventions: Drug: OxyPR followed by OXN PR tablets

INTERVENTIONS:
Drug: OXN PR followed by OxyPR tablets
  Arms: OXN PR followed by OxyPR tablets
Drug: OxyPR followed by OXN PR tablets
  Arms: OxyPR followed by OXN PR tablets

SUMMARY:
The study is intended to explore changes in the composition and quantity of gut bacteria subject to treatment with strong pain medication. Two pain medications will be compared (OXN PR and OxyPR). Other gastrointestinal parameters will be assessed.

DETAILED DESCRIPTION:
Patients who require around-the-clock opioid therapy and show symptoms of constipation secondary to opioid treatment will be randomised to receive either OXN PR followed by OxyPR, or vice versa. Each treatment takes 24days. The study is composed of three phases, a pre-randomisation phase, a double-blind phase and a Follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are receiving WHO step II/III opioid analgesic medication for the treatment of non-malignant pain and who require daily opioid treatment for pain with WHO step III opioid therapy for the duration of the study, based on Investigator's judgement.

Documented history of non-malignant pain that requires around-the-clock opioid therapy (20 - 50 mg oxycodone PR equivalent per day for a minimum of study duration).

Subjects with constipation caused or aggravated by opioids:

* Subject's medical need of regular intake of laxatives to have at least 3 bowel evacuations per week, or having less than 3 bowel evacuations when not taking a laxative.
* In the opinion of the subject and investigator confirm that the subject's constipation is induced, or worsened by the subject's prestudy opioid medication (present at Screening).

Exclusion Criteria:

Any contraindication to oxycodone, naloxone, or any non-investigational medicinal products (NIMPs) that will be used by subjects during the study.

Continuous systemic use of antibiotics and/or steroids within the last 4 weeks prior to the start of the Screening Period and during the study period.

Chronic or intermittent pain that results from Fibromyalgia or Rheumatoid Arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Quantitative analysis of intestinal microbiota as determined in stool samples of subjects treated with OXN PR compared to those treated with OxyPR. As this is an exploratory study, there are no primary objectives, but objectives of main interest. | 8 weeks
  Composition and abundance of selected bacteria in stool samples by means of genomic sequencing of bacterial genes coding for 16S rRNA will be analysed. The analysis will provide information about intra-individual bacterial profile during the study as well as insights about potential effects of treatments, i.e. OXN PR and OxyPR on bacterial profile.
Orocaecal transit time on the basis of intestinal absorption & intermediary bacterial metabolism by breath tests (H2 and CH4 breath test). As this is an exploratory study, there are no primary objectives, but objectives of main interest. | 4 weeks
  Orocaecal time will be measured by H2/CH4/ analysis of expired air of subjects (breath tests). The analysis will provide information about intraindividual changes during the study as well as insights about potential effects of treatments, i.e. OXN PR and OxyPR on orocaecal time.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Gemeinschaftspraxis Loewenstein, Mainz
  - Dr J Hafer, Wetzlar